CLINICAL TRIAL: NCT00876863
Title: A Double-Blind, Placebo-Controlled (Sham Surgery), Randomized, Multicenter Study Evaluating CERE-110 Gene Delivery in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Randomized, Controlled Study Evaluating CERE-110 in Subjects With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Collaborators: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CERE-110-03; NIH Grant 1R01AG030048-01A1
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2017-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Dementia; Memory loss; Cognitive impairment; Nerve growth factor; NGF; Neurotrophic factors; Gene therapy
MeSH Terms: conditions — Alzheimer Disease; Dementia; Memory Disorders; Cognitive Dysfunction; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CERE-110 (Experimental): CERE-110: Adeno-Associated Virus Delivery of NGF
  Interventions: Drug: CERE-110: Adeno-Associated Virus injection Surgery
- Placebo (Sham Comparator): Placebo Surgery
  Interventions: Procedure: Placebo Surgery

INTERVENTIONS:
Drug: CERE-110: Adeno-Associated Virus injection Surgery — Injecting CERE-110 2.0 X 10^11 vg into brain during surgical procedure.
  Arms: CERE-110
Procedure: Placebo Surgery — Placebo Surgery
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the potential benefits of CERE-110 in the treatment of Alzheimer's disease. CERE-110 is an experimental drug that is designed to help nerve cells in the brain function better. CERE-110 uses a virus to transfer a gene that makes Nerve Growth Factor (NGF), a protein that may make nerve cells in the brain healthier and protect them from dying. The virus used in CERE-110 does not cause disease in people. CERE-110 has been carefully studied in laboratory animals and is in the early stages of being tested in people.

Fifty patients with mild to moderate Alzheimer's disease will participate in this study. Half of the study subjects will have CERE-110 injected into the brain during a surgical procedure, while the other half will undergo a "placebo" surgery where no medication will be injected. All study participants will be followed for at least two years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate Alzheimer's disease
* Approved medications for Alzheimer's disease may be taken if the dose has been stable for 3 months
* A study partner who can attend all study visits
* Good general health
* Medically able to undergo neurosurgery

Exclusion Criteria:

* Significant neurological disease other than Alzheimer's disease
* Significant depression or other psychiatric disorder
* Unstable medical conditions

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2015-08-13 (Actual); Study Completion 2015-08-13 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) | 24 Months

SECONDARY OUTCOMES:
Neuropsychological Test Battery | 24 Months
Mini-Mental State Examination (MMSE) | 24 Months
Neuropsychiatric Inventory (NPI) | 24 Months
Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Paul S. Aisen, M.D., Study Director — Alzheimer's Disease Cooperative Study (ADCS)
Locations (10):
- United States (10):
  - University of Alabama, Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Georgetown University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Mount Sinai School of Medicine, New York, New York
  - Duke University, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Medical University of South Carolina, North Charleston, South Carolina
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Rafii MS, Tuszynski MH, Thomas RG, Barba D, Brewer JB, Rissman RA, Siffert J, Aisen PS; AAV2-NGF Study Team. Adeno-Associated Viral Vector (Serotype 2)-Nerve Growth Factor for Patients With Alzheimer Disease: A Randomized Clinical Trial. JAMA Neurol. 2018 Jul 1;75(7):834-841. doi: 10.1001/jamaneurol.2018.0233. PMID 29582053